CLINICAL TRIAL: NCT04994665
Title: Evaluation of Omentopexy on Gastro-oesophageal Reflux Following Sleeve Gastrectomy
Acronym: Sleevepexie
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHD21_0032
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: sleeve gastrectomy; omentopexy; gastro-oesophageal disease
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve gastrectomy (Active Comparator): realization of a sleeve gastrectomy alone
  Interventions: Procedure: sleeve gastrectomy
- sleeve gastrectomy with omentopexy (Experimental): realization of a sleeve gastrectomy followed by an omentopexy
  Interventions: Procedure: sleeve gastrectomy with omentopexy

INTERVENTIONS:
Procedure: sleeve gastrectomy — The sleeve gastrectomy is a surgical weight-loss procedure, about 80% of the stomach is removed
  Arms: Sleeve gastrectomy
Procedure: sleeve gastrectomy with omentopexy — After sleeve gastrectomy procedure, the omentopexy involves suturing the omentum back to the greater curvature of the stomach in several locations, depending on the length of the greater curvature
  Arms: sleeve gastrectomy with omentopexy

SUMMARY:
The aim of the study is to assess impact of omentopexy on de novo gastro-oesophageal reflux disease (GERD) after sleeve gastrectomy.

This will be assess 2 years postoperatively. This study is a prospective, multicentric, randomized trial. Five hundred twenty six patients should be included with 263 in each arm. First arm will include patients who have a sleeve gastrectomy. The second arm will include patients who have sleeve gastrectomy with omentopexy.

Two years after surgery , it will be collected a CARLSSON score and BAROS score (quality of life).

The main objective is to show that omentopexy decreases the rate of de novo GERD after sleeve gastrectomy at 2 years postoperatively without the use of Proton-Pump Inhibitors (PPIs)

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* Patient to be operated in first intention of a sleeve gastrectomy
* Initial BMI between 35Kg/m² and 40 Kg/m² associated with at least one severe comorbidity likely to be improved after surgery according to HAS recommendations.

OR initial BMI ≥ 40 Kg/m².

* Multidisciplinary follow-up of at least 6 months before surgery
* Validation of the surgical intervention in a multidisciplinary consultation meeting
* Certificate of no contraindication by a psychiatrist
* Patient who has the capacity to understand the protocol and has given consent to participate in the research,
* Patient with social security coverage.

Exclusion Criteria:

* Eating disorder or mental disorder
* Misunderstanding of the protocol
* Psychiatric contraindication
* Initial BMI <35Kg/m².
* Initial BMI between 35Kg/m² and 40 Kg/m² without comorbidities.
* Esophagitis of grade B and above on the Oeso-Gastro-Duodenal Fibroscopy
* CARLSSON score (score ≥ 4) preoperatively
* Presence of a Proton-Pump Inhibitors treatment
* Patient to have a 2-stage surgery (first sleeve gastrectomy then gastric bypass or Single Anastomosis Duodeno-Ileal bypass)
* Patient participating in another interventional clinical research protocol involving a drug or medical device
* Patient who are pregnant, breastfeeding, or who have the potential to become pregnant without effective contraception at the time of inclusion and up to 24 months after surgery
* Patient under guardianship, curators or legal protection,P

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate de novo GERD of patient benefited from sleeve gastrectomy with omentopexy versus sleeve gastrectomy alone | 2 years postoperatively
  Presence of de novo GERD defined by a clinical score of CARLSSON >= 4 and/or the use of a PPIs treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emeric Abet, Dr, Principal Investigator — CHD Vendée
Locations (9):
- France (9):
  - CH de la Cote Basque, Bayonne
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - CHU Nantes, Nantes
  - Clinique Jules Verne, Nantes
  - Centre Hospitalier Régional et Universitaire d'Orléans, Orléans
  - Hopital Pontchaillou, Rennes
  - Clinique Mutualiste de la Sagesse, Rennes
  - Clinique Santé Atlantique, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No